CLINICAL TRIAL: NCT03654716
Title: Phase 1 Study of the Dual MDM2/MDMX Inhibitor ALRN-6924 in Pediatric Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: TeamConnor Childhood Cancer Foundation (Unknown); Cookies for Kids' Cancer (Other); Aileron Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, David S Shulman, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-284
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Leukemia; Brain Tumor; Solid Tumor; Lymphoma
Keywords: Leukemia; Solid Tumor; Brain Tumor; Lymphoma; TP53; p53; MDM2; MDMX; PPM1D
MeSH Terms: conditions — Leukemia; Brain Neoplasms; Lymphoma | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ALRN-6924 -- Cohort A (Experimental): * Participants will receive ALRN-6924 monotherapy on days 1, 4 (± 1 day), 8 (± 1 day), and 11 (± 1 day) of a 21-day cycle.
  * ALRN-6924 will be administered intravenously.
  * Participants with otherwise unselected TP53 wild type solid tumors and lymphoma will participate in this cohort.
  Interventions: Drug: ALRN-6924
- ALRN-6924 -- Cohort B (Experimental): * Participants will receive ALRN-6924 monotherapy on days 1, 4 (± 1 day), 8 (± 1 day), and 11 (± 1 day) of a 21-day cycle.
  * ALRN-6924 will be administered intravenously.
  * Participants with solid and CNS tumors and lymphoma with specific diagnoses or molecular features will participate in this cohort.
  Interventions: Drug: ALRN-6924
- ALRN-6924 -- Cohort C (Experimental): * Patients will receive ALRN-6924 in combination with cytarabine on days 1, 8 (± 1 day), and 15 (± 1 day) of a 28-day cycle.
  * Cytarabine is administered intravenously.
  * ALRN-6924 will be administered intravenously.
  * Participants with TP53 wild type acute leukemia will participate in this cohort.
  Interventions: Drug: ALRN-6924; Drug: Cytarabine

INTERVENTIONS:
Drug: ALRN-6924 — ALRN-6924 is a drug that blocks certain proteins in tumor cells called MDM2 and MDMX. These proteins may be important in the growth of some cancers. Laboratory experiments and results from studies with adults show that ALRN-6924 may stop tumor growth and, in some cases, may cause tumor cells to die.
Drug: Cytarabine — Cytarabine belongs to the category of chemotherapy called antimetabolites. Antimetabolites are very similar to normal substances within the cell. When the cells incorporate these substances into the cellular metabolism, they are unable to divide
  Other Names: Cytosar
  Arms: ALRN-6924 -- Cohort C

SUMMARY:
This research study is studying a novel drug called ALRN-6924 as a possible treatment for resistant (refractory) solid tumor, brain tumor, lymphoma or leukemia.

The drugs involved in this study are:

* ALRN-6924
* Cytarabine (for patients with leukemia only)

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied.

In this research study, the investigators are evaluating a new drug, ALRN-6924, as a potential new treatment for children with cancer.

The FDA (the U.S. Food and Drug Administration) has not approved ALRN-6924 as a treatment for any disease.

This is the first time that ALRN-6924 will be studied in children.

ALRN-6924 is a drug that blocks certain proteins in tumor cells called MDM2 and MDMX. These proteins may be important in the growth of some cancers. Laboratory experiments and results from studies with adults show that ALRN-6924 may stop tumor growth and, in some cases, may cause tumor cells to die. ALRN-6924 has been tested in adults with cancer to find out about side effects and dosing in adults.

The purposes of this study are:

* to evaluate side effects of ALRN-6924 and to find the best dose of ALRN-6924 when used in children.
* to determine whether this drug may have benefits against the types of cancer seen in children
* to see how the body breaks down ALRN-6924 by measuring the amount of ALRN-6924 in the blood.

One part of the study is for children with solid tumors, lymphoma, and brain tumors (Cohorts A or B). Another part of this study is for children with leukemia (Cohort C).

ELIGIBILITY:
Inclusion Criteria:

* Age > 1 years and ≤ 21 years at time of enrollment.
* Karnofsky performance status ≥ 50% for patients ≥16 years of age and/or Lansky ≥ 50% for patients <16 years of age
* For Cohorts A and B

  * Participants must have evaluable or measurable disease.
  * Must have disease that is relapsed or refractory and for which standard curative or palliative measures do not exist or are no longer effective.
  * For Cohort A, participants must have histologically confirmed non-CNS primary solid tumors or lymphoma based upon biopsy or surgery at initial diagnosis and/or relapse/progression. The only exception to histologic confirmation is for patients with retinoblastoma.
  * For Cohort B, participants must have one of the following confirmed diagnoses:

    * Diagnosis of retinoblastoma
    * Histologic diagnosis of hepatoblastoma and WT TP53
    * Diagnosis of malignant rhabdoid tumor and WT TP53. For the purposes of this study, a diagnosis of malignant rhabdoid tumor will include histologic diagnosis (CNS atypical teratoid/rhabdoid tumor, rhabdoid tumor of the kidney or rhabdoid tumor of the soft tissue) AND molecular confirmation (loss of INI1 protein staining or BRG1 protein staining by IHC, or documentation of SMARCB1 or SMARCA4 mutation or loss)
    * Solid tumor, CNS tumor, or lymphoma with MDM2 amplification or high-copy gain and WT TP53
    * Solid tumor, CNS tumor, or lymphoma with MDMX amplification or high-copy gain and WT TP53
    * Solid tumor, CNS tumor, or lymphoma with PPM1D amplification, high-copy gain, or PPM1D activating mutation and WT TP53
    * Solid tumor or lymphoma with TET2 loss or loss-of-function mutation and WT TP53
    * Testing for MDM2, MDMX, TP53, SMARCB1, SMARCA4, PPM1D and TET2 variants must be performed in a laboratory certified to return results for clinical purposes in order to be used to qualify a patient for Cohort B.
* For Cohort C

  * Participants must have a histologically confirmed diagnosis of relapsed or refractory AML, ALL, mixed lineage leukemia, biphenotypic leukemia, or other undifferentiated acute leukemia with one of these disease states:
  * Refractory disease defined as: Persistent disease after at least two induction cycles; OR
  * Relapsed disease defined as: Second or subsequent relapse, or any relapse that is refractory to salvage chemotherapy
  * Subjects in Cohort C must have ≥ 5% blasts (M2 or M3 marrow) definitively identified either on a bone marrow aspirate or biopsy sample, as assessed by morphology, immunohistochemical studies, flow cytometry, karyotype, cytogenetic testing such as fluorescent in situ hybridization (FISH) or other molecular studies.
  * Subjects must have CNS1 or CNS2 disease.
* Absence of inactivating TP53 alteration by Next Generation Sequencing assay or PCR-based assay in a laboratory certified to return results for clinical purposes.
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy except organ function as noted below. Patients must meet the following minimum washout periods prior to enrollment:
* Myelosuppressive chemotherapy: At least 14 days after the last dose of myelosuppressive chemotherapy (42 days for nitrosourea or mitomycin C).

Patients on Cohort C may have received any of the following medications without a "wash-out" period as long as other organ function requirements are met (methotrexate must not be given within 48 hours of ALRN-6924 planned start):

Standard maintenance therapy [any combination of vincristine, 6-mercaptopurine, corticosteroids, and/or low-dose methotrexate (45 mg/m2/week or less)]; Hydroxyurea; Patients on any cohort may have received intrathecal chemotherapy with methotrexate, hydrocortisone and/or cytarabine (non-liposomal) without a "wash-out" period as long as other organ function requirements are met (methotrexate must not be given within 48 hours of ALRN-6924 planned start).

* Radiotherapy:

  * At least 14 days after local XRT (small port, including cranial radiation);
  * At least 90 days must have elapsed after prior TBI, craniospinal XRT or if >50% radiation of pelvis;
  * At least 42 days must have elapsed if other substantial BM radiation;
  * At least 42 days must have passed since last MIBG or other radionuclide therapy.
* Small molecule biologic therapy: At least 7 days following the last dose of a biologic agent. For agents with known adverse events occurring beyond 7 days, this duration must be extended beyond the time in which adverse events are known to occur. If extended duration is required, this should be discussed with and approved by the overall PI.
* Monoclonal antibody: At least 21 days must have elapsed after the last dose of antibody.
* Myeloid growth factors: At least 14 days following the last dose of long-acting growth factor (e.g. Neulasta) or 7 days following short-acting growth factor.
* Autologous hematopoietic stem cell transplant and stem cell boost: Patients must be at least 60 days from day 0 of an autologous stem cell transplant or stem cell boost.
* Allogeneic hematopoietic stem cell transplant or cellular therapies (including CAR-T cells): The patient must have no evidence of graft versus host diseaseand at least 90 days must have elapsed after allogeneic stem cell infusion. At least 42 days must have elapsed after last dose of other cellular therapy.
* Solid Organ Transplantation: Patients with hepatoblastoma treated with liver transplantation will be eligible to enroll if they meet all of the following requirements:

  * At least 90 days must have elapsed from the date of liver transplant;
  * No clinical or radiographic evidence of rejection since the date of transplant; AND
  * All organ function requirements are met.
* Major Surgery: At least 2 weeks from prior major surgical procedure. Note: Biopsy, CNS shunt placement/revision, and central line placement/removal are not considered major.
* MDM2 inhibitors: Patients for Cohorts A and C may have received prior MDM2 inhibitor therapy. Patients in Cohort B must not have received prior MDM2 inhibitor therapy. Patients in all cohorts must not have received dual MDM2/MDMX inhibition.
* Participants must have normal organ function as defined below.
* Bone Marrow Function for Subjects in Cohorts A and B without Bone Marrow Involvement by Disease:

  * Absolute neutrophil count ≥1,000 /uL
  * Platelets ≥75,000 /uL and transfusion independent, defined as not receiving a platelet transfusion for at least 5 days prior to CBC documenting eligibility.
* Hematologic Requirements for Subjects in Cohorts A and B with Bone Marrow Involvement by Disease:

  * Absolute neutrophil count ≥750 /uL
  * Platelets ≥50,000 /uL (may receive platelet transfusions)
  * Not known to be refractory to red cell and/or platelet transfusions.
* Bone Marrow Function for Subjects in Cohorts C with Acute Leukemia

  ---Not known to be refractory to red cell and/or platelet transfusions
* Hepatic Function:

  * Total bilirubin ≤ 1.5 x upper limit of normal for age except for patients with known Gilbert syndrome who may enroll using direct bilirubin ≤ 1.5 x upper limit of normal for age as bilirubin criterion
  * ALT (SGPT) ≤ 3 x upper limit of normal (135 U/L). For the purpose of this study, the ULN for ALT is 45 U/L. Patients with acute leukemia AND leukemic infiltration of the liver may enroll to Cohort C if ALT < grade 2 and total bilirubin meets above requirement.
  * Serum albumin > 2 g/dL
* Renal Function:

  * A serum creatinine within protocol limits based on age/sex. OR
  * Creatinine clearance ≥ 60 mL/min/1.73 m2 for participants with creatinine levels greater than the above age/sex maximum allowed values.
* Adequate Cardiac Function: QTc < 480 msec
* For patients with CNS tumors (primary or metastatic), any baseline neurologic deficits (including seizure) must be stable for at least one week prior to study enrollment. Patients with CNS tumors receiving corticosteroids must be on a stable or decreasing dose at time of study entry.
* Ability to understand and/or the willingness of the patient (or parent or legally authorized representative, if minor) to provide informed consent, using an institutionally approved informed consent procedure.
* Participants of child-bearing or child-fathering potential must agree to use adequate contraception (hormonal birth control; intrauterine device; double barrier method; or total abstinence) throughout their participation, including up until 30 days after last dose of ALRN-6924.

Exclusion Criteria:

* Patients receiving medications within 48 hours of enrollment that are primarily cleared by organic anion transporter polypeptide [OATP] members OATP1B1 and OATP1B3
* Pregnant participants will not be entered on this study given that the effects of ALRN-6924 on the developing human fetus are unknown.
* Breastfeeding mothers are not eligible, because there is an unknown risk for adverse events in nursing infants secondary to treatment of the mother with ALRN-6924.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ALRN-6924.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with a known history of HIV, hepatitis B, and/or hepatitis C (testing not required as part of screening).
* Patients with a known personal history of angioedema or known family history of hereditary angioedema.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with dose limiting toxicity by CTCAE v.5.0 for each dose level | 2 years
Percentage of patients with toxicity by CTCAE v.5.0 | 2 Years

SECONDARY OUTCOMES:
Peak plasma concentration of ALRN-6924 | 2 years
Area under the curve (AUC) of ALRN-6924 | 2 years
Objective response rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David S Shulman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No